CLINICAL TRIAL: NCT01374711
Title: The Effects of Immunostimulation With GM-CSF or IFN-y on Immunoparalysis Following Human Endotoxemia. A Parallel Randomized Double-blind Placebo-controlled Study
Brief Title: The Effects of Immunostimulation With GM-CSF or IFN-y on Immunoparalysis Following Human Endotoxemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Peter Pickkers, MD, PhD, Radboud University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NL36068.091.11 BI
Record Dates: First submitted 2011-05-19; First posted 2011-06-16 (Estimated); Last update posted 2013-06-27 (Estimated); Status verified 2013-06

CONDITIONS: Endotoxemia; Inflammation; Multi Organ Dysfunction Syndrome; Sepsis
Keywords: Endotoxin; Inflammation; Sepsis; GM-CSF; IFN-y
MeSH Terms: conditions — Endotoxemia; Inflammation; Sepsis | interventions — Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- placebo (Placebo Comparator): LPS will be administered twice on days 1 and 7. In between placebo will be administered on days 2, 4 and 6 subcutaneously.
  Interventions: Other: E.coli endotoxin
- GM-CSF (Active Comparator): LPS will be administered twice on days 1 and 7. In between GM-CSF will be administered on days 2, 4 and 6 subcutaneously.
  Interventions: Drug: GM-CSF; Other: E.coli endotoxin
- IFN-y (Active Comparator): LPS will be administered twice on days 1 and 7. In between IFN-Y will be administered on days 2, 4 and 6 subcutaneously.
  Interventions: Drug: IFN-Y; Other: E.coli endotoxin

INTERVENTIONS:
Drug: GM-CSF — GM-CSF (4microgram/kg/day subcutaneously) on days 2, 4 and 6.
  Arms: GM-CSF
Drug: IFN-Y — IFN-Y (100 microgram/day, subcutaneously) on days 2, 4 and 6.
  Arms: IFN-y
Other: E.coli endotoxin — 2 ng/kg E.coli reference endotoxin 11:H 10:K negative intravenously

SUMMARY:
The human body knows a biphasic immunological reaction to sepsis. First, the pro-inflammatory reaction takes place, marked by the release of pro-inflammatory cytokines like TNF-α, as a reaction to the bacterial toxins. Secondly, the counter regulatory anti-inflammatory reaction arises. This phase is acting as negative feedback on the inflammation by inhibition of the pro-inflammatory cytokines. This is called "immunoparalysis", a pronounced immunosuppressive state, which renders patients vulnerable to opportunistic infections. Most of the septic patients survive the initial pro-inflammatory phase, but die during this second stage.Research in the past has shown that immunostimulatory therapy with GM-CSF or IFN-γ has promising effects on the pro-inflammatory reaction during immunoparalysis ex vivo. Both drugs are known for their immunostimulatory effects. Recent pilot studies have showed in septic patients, that long-lasting monocyte deactivation in sepsis ex vivo can be reversed by these two immunostimulants. However, the mechanism and extent of immunoparalysis recovery may be different between the two compounds. Previously it has been shown that human endotoxemia (induced by LPS), leads to marked immunosuppression in healthy individuals, characterized by a transient refractory state to a subsequent LPS challenge (endotoxin tolerance). Consequently, human endotoxemia can serve as a standardized, controlled model for sepsis-induced immunoparalysis. Until now, all studies have focused on the ex vivo tolerance. However, we have recently proved, that the ex vivo condition is not completely representative for the in vivo situation. Ex vivo, leukocyte tolerance to LPS resolves within one day, while the in vivo immunoparalysis persists for two weeks. In this project, we will investigate the effects of both GM-CSF and IFN-γ in a parallel double-blind placebo controlled randomized manner on the immunoparalysis following human endotoxemia, both in-vitro and in vivo. As a result, we hope to get more insight in the pathophysiology of sepsis-induced immunoparalysis and thereby develop new immunostimulatory therapies that improve patient outcome

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers

Exclusion Criteria:

* seropositivity for markers of hepatitis B or HIV infection or medical history of any other obvious disease associated with immune deficiency
* Use of any medication or drugs
* a history of adverse reaction or hypersensitivity to GM-CSF/ IFN-γ
* Smoking.
* Previous spontaneous vagal collapse.
* History, signs or symptoms of cardiovascular disease.
* (Family) history of myocardial infarction or stroke under the age of 65 years.
* Cardiac conduction abnormalities on the ECG consisting of a 2nd degree atrioventricular block or a complex bundle branch block.
* Hypertension (defined as RR systolic > 160 or RR diastolic > 90) or hypotension (defined as RR systolic < 100 or RR diastolic < 50).
* Renal impairment (defined as plasma creatinin >120 μmol/l).
* Liver enzyme abnormalities or positive hepatitis serology.
* Febrile illness during the week before the LPS challenge
* Participation in a drug trial or donation of blood 3 months prior to the LPS challenge.
* Chronic hiccups (defined as hiccups longer than 15 minutes in the past 6 months)
* Pre-existent muscle disease (congenital or acquired) or diseases / disorders know to be associated with myopathy including diabetes and auto-immune diseases.
* Pre-existent lung disease
* Upper airway / esophageal pathology
* Recent (< 1 month) nasal bleeding
* Phrenic nerve lesions
* Any metals in body (pacemaker, splinters, metal stitches)

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2011-05; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
the effects of GM-CSF/IFN-γ on the development of in vivo immunoparalysis induced by experimental human endotoxemia | 1 week (day 1- day 8)
  This will be determined by measuring plasma levels of various pro and anti-inflammatory cytokines and assessing the difference in the LPS-induced cytokine response between day 1 and 7

SECONDARY OUTCOMES:
The effects of GM-CSF/IFN-γ on the ex-vivo responsiveness of leukocytes to various inflammatory stimuli | 1 week (day 1- day 8)
the effects of GM-CSF/IFN-γ on monocyte HLA-DR expression | 1 week (day 1- day 8)
the effects of GM-CSF/IFN-γ on transcriptional pathways of leukocytes (qPCR and microarray) | 1 week (day 1- day 8)
the effects of GM-CSF/IFN-γ on urine markers of tubular injury | 1 week (day 1- day 8)
The effect of LPS on twitch transdiaphragmatic pressure | 1 day
the effects of GM-CSF/IFN-γ on clinical symptoms (illness score, mean arterial pressure, heart rate and temperature) | 1 week (day 1- day 8)
the effects of GM-CSF/IFN-γ on changes in phenotype and gene expression caused by mechanisms other than changes in the underlying DNA sequence | 1 week (day 1- day 8)
Beta 2 Glycoprotein and platelet-monocyte interactions post-LPS | 1 day
Macrophage differentiation | 1 day
Immunosuppressive neutrophil populations | 1 week (day 1- day 8)
Blood viscosity | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Peter Pickkers, Prof, MD, PhD, Principal Investigator — Radboud University Nijmegen Medical Centre, The Netherlands
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Derived] Leentjens J, Kox M, Koch RM, Preijers F, Joosten LA, van der Hoeven JG, Netea MG, Pickkers P. Reversal of immunoparalysis in humans in vivo: a double-blind, placebo-controlled, randomized pilot study. Am J Respir Crit Care Med. 2012 Nov 1;186(9):838-45. doi: 10.1164/rccm.201204-0645OC. Epub 2012 Jul 19. PMID 22822024